CLINICAL TRIAL: NCT03722732
Title: Comparison of Blood Loss in Laparoscopic vs Open Pancreaticoduodenectomy in Patients With Periampullary Carcinoma - A Randomized Clinical Trial
Brief Title: Comparison of Blood Loss in Laparoscopic vs Open Pancreaticoduodenectomy in Patients With Periampullary Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Principal Investigator, Hirdaya H Nag, MS, Professor, Govind Ballabh Pant Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.1/IEC/MAMC/63/03/18/NO325
Record Dates: First submitted 2018-10-02; First posted 2018-10-29 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Periampullary Carcinoma
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open pancreaticoduedenectomy (Active Comparator): will include all the patients who will undergo open pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy
- Laparoscopic pancreaticoduodenectomy (Active Comparator): will include all the patients undergoing laparoscopic pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — pancreaticoduodenectomy either laparoscopically or open will be done

SUMMARY:
the study is designed to compare the blood loss between laparoscopic vs open pancreaticoduodenectomy in a randomized clinical trial

DETAILED DESCRIPTION:
the study will assess the difference in the amount of blood loss in Lap vs Open WPD. the amount of blood loss will be calculated on the basis of a formula which takes pre operative and post operative hematocrit, PCV and blood volume into consideration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both the sex aged between >18 years.
2. Patients with a diagnosis of resectable periampullary carcinoma on imaging.
3. Patients with ASA grade 1 or 2

Exclusion Criteria:

* 1) Patients found to have unresectable disease on radiological investigation. 2) Patients with ASA grade 3 or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss in ml, quantitative | 24 hours
  blood loss will be assessed with the help of a formula which uses preoperative and post operative hematocrit, blood volume and PCV

CONTACTS AND LOCATIONS:
Overall Officials: H H Nag, MS, Principal Investigator — GBPant Hospital
Locations (1):
- G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No